CLINICAL TRIAL: NCT02695069
Title: Random Placenta Margin Incision for Hemorrhage Control During Cesarean Section of Complete Placenta Previa Pregnancies
Brief Title: Efficacy Study of Random Placenta Margin Incision to Treat Complete Placenta Previa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhengping Liu, MD, Director, Maternal and Child Health Hospital of Foshan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCHHFoshan-1601
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Complete Placenta Previa
Keywords: Complete Placenta Previa; Random Placenta Margin Incision; Cesarean Section; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Participants (Experimental): A random hysterotomy incision is done in the placenta margin. To precisely determine the placental location and the edge of the placenta, preoperative ultrasonography is used in determining the optimal place for the uterine incision.
  Interventions: Procedure: Random Placenta Margin Incision

INTERVENTIONS:
Procedure: Random Placenta Margin Incision — A random hysterotomy incision is done in the placenta margin. To precisely determine the placental location and the edge of the placenta, preoperative ultrasonography is used in determining the optimal place for the uterine incision.

SUMMARY:
The purpose of this study is to assess the efficacy of random placenta margin incision for hemorrhage control during cesarean section of complete placenta previa pregnancies.

DETAILED DESCRIPTION:
Placenta previa is used to describe a placenta that is implanted over or very near the internal cervical os and the complete placenta previa is defined that the internal os is covered completely by placenta. This obstetric complication is associated with high risks for maternal hemorrhage and emergency peripartum hysterectomy can be the only effective action to take, although it carries many morbidities for the women especially those with low parity. Although, nowadays the obstetrician can diagnose placenta previa before delivery, it is still one of the important causes of maternal mortality. The only safe and appropriate mode of delivery for placenta previa is by cesarean delivery. In the absence of accreta, this can usually be accomplished using a lower segment uterine incision. Because of cutting through the placenta, it is often associated with increased maternal bleeding. In addition, the umbilical cord will be also excessive blood loss when the placenta is transected. Theoretically, random placenta margin incision can effectively avoid the damage of the placenta and reduce the maternal blood loss.

The investigators conduct a prospective study to assess the efficacy of random placenta margin incision for hemorrhage control during cesarean section of complete placenta previa pregnancies at Department of Obstetrics, Southern Medical University Affiliated Maternal and Child Health Hospital of Foshan, since January 2016 till December 2016, after approval of the study protocol by the Local Ethical Committee.

All participants have complete placenta previa and provide written informed consent to undergo any procedure necessary as an attempt to avoid hysterectomy. And they also provide written informed consent to undergo hysterectomy if all measures attempted to preserve the uterus fail.

To precisely determine the placental location and the edge of the placenta, preoperative ultrasonography is used in determining the optimal place for the uterine incision. The investigator performed all cesarean deliveries and assisted by the second investigator. The parietal peritoneum is opened by sharp dissection and blunt expansion, if necessary, high above the bladder, a bladder flap is made and the bladder is retracted. A random hysterotomy incision is done in the placenta margin. It is expanded on both sides using scissors, stopping shortly before the uterine arteries. Active delivery of the placenta is attempted by searching manually for a plane of cleavage between the placenta and the uterus after delivery of the fetus. In addition to uterotonics, measures such as "oversewing" of the placental bed, intrauterine balloon tamponade, and B-Lynch or other compression sutures are also used depending on different circumstances.

ELIGIBILITY:
Inclusion Criteria:

* A gestation age of ≥ 28 weeks
* Delivered by cesarean section
* Antepartum diagnosis of complete placenta accreta by obstetric ultrasound and doppler

Exclusion Criteria:

* Women who refuse to participate
* Pregnant women with serious diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Postpartum Hemorrhage | within the first 30 days after cesarean section

SECONDARY OUTCOMES:
Number of blood products transfused | within the first 30 days after cesarean section
Length of hospitalization | 6 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Zhengping Liu, MD, Principal Investigator — Maternal and Child Health Hospital of Foshan
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided